CLINICAL TRIAL: NCT02092064
Title: Association Between Basal Proteinuria Levels and Pregnancy Outcomes in Familial Mediterranean Fever
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, cantekin iskender, Perinatology, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: Basal Proteinuria in FMF
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Basal Proteinuria in Pregnancy
Keywords: basal proteinuria; FMF; pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Biospecimen Retention: None Retained — maternal ürine protein level
Oversight: Data Monitoring Committee: No

SUMMARY:
to investigate the effect of basal proteinuria on pregnancy outcomes of patients with Familial Mediterranean fever (FMF).

DETAILED DESCRIPTION:
Familial Mediterranean fever (FMF) is also known recurrent polyserositis the most common hereditary recurrent febrile disorder. It is characterized by paroxysmal episodes of the high fever and signs of serositis-peritonitis, pleuritis, synovitis. Between these attacks, patients are usually asymptomatic. FMF mainly affects populations of the Mediterranean region such as Turks.

The diagnosis of FMF may be extremely difficult to establish in the presence of atypical signs, and absence of family history . Colchicine is effective in most of the patients with FMF. The one the most important complications of FMF is the development of renal amyloidosis. It potentially progress sequentially through preclinical, proteinuric, nephrotic, azotemic and uremic stages to end stage renal disease if not treated properly with colchicine. Previous studies suggests that colchicine does not appear to be a major human teratogen, and, probably, has no cytogenetic effect.

FMF affects females mainly in their childbearing years. FMF is associated with higher rates of recurrent abortion, premature rupture of membranes (PROM) and preterm birth. Despite of adverse outcomes have been reported in pregnants with FMF the outcome of pregnancies in FMF appear favorable with the healthy population since the usingof the colchicine. Although the effect of pregnancy on the course of FMF related amyloidosis is controversial, it is generally accepted that renal function may disrupt during pregnancy.

Few studies have investigated the effect of FMF complications (amyloidosis and nephrotic syndrome) on pregnancy course.

The aim of this study is to investigate the effect of basal proteinuria on pregnancy outcome of patients with Familial Mediterranean fever (FMF).

ELIGIBILITY:
Inclusion Criteria:

* pregnant patients with FMF

Exclusion Criteria:

* multiple pregnancies

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant patients with FMF
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-10 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
change in proteinuria correlation to the adverse outcomes of pregnancy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: dilek uygur, Principal Investigator — zekai tahir burak hospital
Locations (1):
- Zekai Tahir Burak Maternity Hospital, Ankara, Altindag, Turkey (Türkiye)

REFERENCES:
- [Result] Turgal M, Selcuk I, Ozyuncu O. Pregnancy outcome of five patients with renal amyloidosis regarding familial Mediterranean fever. Ren Fail. 2014 Mar;36(2):306-8. doi: 10.3109/0886022X.2013.846863. Epub 2013 Oct 29. PMID 24168456
- [Result] Yasar O, Iskender C, Kaymak O, Taflan Yaman S, Uygur D, Danisman N. Retrospective evaluation of pregnancy outcomes in women with familial Mediterranean fever. J Matern Fetal Neonatal Med. 2014 May;27(7):733-6. doi: 10.3109/14767058.2013.837446. Epub 2013 Sep 25. PMID 23981183